CLINICAL TRIAL: NCT03108911
Title: Gluten Free Diet for AML Patients Undergoing Induction Chemotherapy
Brief Title: Gluten Free Diet in Diminishing Side Effects Patients With Acute Myeloid Leukemia Undergoing Induction Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: limited resources
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 021702; NCI-2017-00498 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 021702 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH)
Record Dates: First submitted 2017-04-06; First posted 2017-04-11 (Actual); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Practice Guidelines as Topic; Standard of Care; Diet Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (GFD) (Experimental): Patients receive GFD prepared by the hospital per dietary/nutrition pharmacy standards from the initiation of induction chemotherapy until hospital discharge (approximately 30 days). Patients also complete a daily food intake diary. A stool sample is collected from patients at baseline, day 14, and on the day of hospital discharge for gut microbiome analysis.
  Interventions: Procedure: Biospecimen Collection; Other: Dietary Intervention; Other: Laboratory Biomarker Analysis
- Group II (standard diet) (Experimental): Patients receive a standard diet for from the initiation of induction chemotherapy until hospital discharge (approximately 30 days). Patients also complete a daily food intake diary. A stool sample is collected from patients at baseline, day 14, and on the day of hospital discharge for gut microbiome analysis.
  Interventions: Other: Best Practice; Procedure: Biospecimen Collection; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Best Practice — Receive standard diet
  Other Names: standard of care; standard therapy
  Arms: Group II (standard diet)
Procedure: Biospecimen Collection — Provide stool sample
Other: Dietary Intervention — Receive GFD
  Other Names: Dietary Modification; intervention, dietary; Nutrition Intervention; Nutrition Interventions; Nutritional Interventions
  Arms: Group I (GFD)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized phase II trial studies how well a gluten free diet works in diminishing side effects in patients with acute myeloid leukemia undergoing induction chemotherapy. A gluten free diet may result in less intestinal side effects and blood infections during the induction chemotherapy compared to a standard diet.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if a gluten free diet (GFD) modulates the rate and severity of bacteremia and gastrointestinal toxicity (measured by total parenteral nutrition [TPN] or nothing by mouth [NPO] order) in patients undergoing standard acute myeloid leukemia (AML) induction chemotherapy.

SECONDARY OBJECTIVES:

I. To determine the tolerance of, and compliance with, a GFD in patients undergoing standard AML induction chemotherapy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients receive GFD prepared by the hospital per dietary/nutrition pharmacy standards from the initiation of induction chemotherapy until hospital discharge (approximately 30 days). Patients also complete a daily food intake diary. A stool sample is collected from patients at baseline, day 14, and on the day of hospital discharge for gut microbiome analysis.

GROUP II: Patients receive a standard diet for from the initiation of induction chemotherapy until hospital discharge (approximately 30 days). Patients also complete a daily food intake diary. A stool sample is collected from patients at baseline, day 14, and on the day of hospital discharge for gut microbiome analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing AML induction chemotherapy with an anthracycline + cytarabine-based chemotherapy regimen
* No history of celiac disease or non-celiac gluten sensitivity
* No grade 3 or 4 gastrointestinal (GI) toxicity at time of initial screening
* No documented bacteremia at time of initial screening
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2 at time of initial screening

Exclusion Criteria:

* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-07-27 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

PRIMARY OUTCOMES:
Rate and severity of bacteremia with enteric organisms during AML induction therapy assessed using stool samples | Up to 30 days
  To determine how often patients develop bacteremia during AML induction therapy
Rate and severity of GI symptoms during AML induction therapy | Up to 30 days
  To determine what the severity is if GI symptoms develops
Rate of compliance with GFD assessed using daily food intake diary | Up to 30 days
  Adherence to diet will be recorded in a food diary. Compliance will be defined as > 67% of meals being gluten free.

CONTACTS AND LOCATIONS:
Overall Officials: Roger Strair, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (1):
- Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey, United States